CLINICAL TRIAL: NCT04753996
Title: Characterization of Biliary Cell-derived Organoids from Bile of PSC and Non-PSC Patients
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-012867; RC2DK118619 (NIH)
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Primary Sclerosing Cholangitis; PSC; Cholangiocarcinoma
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of bile and biliary brushings collected at time of endoscopic retrograde cholangiopancreatography (ERCP) or cholecystectomy (gallbladder removal).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Sclerosing Cholangitis (PSC): Subjects diagnosed with Primary Sclerosing Cholangitis (PSC) will be asked to provide bile and/or brush cytology at time of endoscopic retrograde cholangiopancreatography (ERCP) or cholecystectomy (gallbladder removal).
- Control (non-PSC): Subjects without a diagnosis of Primary Sclerosing Cholangitis (PSC) will be asked to provide bile and/or brush cytology at time of endoscopic retrograde cholangiopancreatography (ERCP) or cholecystectomy (gallbladder removal).

SUMMARY:
The purpose of this research is to create a collection of bile, bile duct brushings and medical information from people with Primary Sclerosing Cholangitis (PSC) and controls to learn more about changes that occur in the liver.

DETAILED DESCRIPTION:
The study will ask participants to provide bile and/or bile duct cytology brushings at time of endoscopic retrograde cholangiopancreatography (ERCP) or cholecystectomy (gallbladder removal). The bile and brushings will be used to generate and perpetuate bile-derived organoids using an established matrigel-based protocol. These organoids will then be used in downstream experiments to better understand disease-specific alterations to biological pathways informative of disease pathogenesis

ELIGIBILITY:
Inclusion Criteria:

PSC

* Patients diagnosed with PSC between the age of 18 and 85.
* The diagnosis of PSC will be based on standard PSC criteria including clinical and biochemical evidence of chronic cholestasis of at least six months duration, positive cholangiographic findings and compatible liver biopsies if available.
* Women with PSC of childbearing potential and pregnant women will be offered enrollment because there is no risk to an unborn child in this investigation. Patients with PSC and Cholangiocarcinoma will be included.

Controls

• Controls without history of PSC or evidence of other chronic liver disease of either gender that will participate in this study should be between the ages of 18-85.

Exclusion Criteria:

* Patients unable to provide inform consent.
* Prisoners and institutionalized individuals.
* PSC with orthotopic liver transplantation
* History of Roux En Y procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Primary Sclerosing Cholangitis (PSC) and controls without PSC will be able to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants in study. | 20 years
  Number of participants in study.

SECONDARY OUTCOMES:
Number of samples (per type) | 20 years
  Number of samples collected (bile liquid, biliary cells)
Number of clinical phenotypes and/or observations. | 20 years
  Number of clinical phenotypes and/or endpoints observed (i.e. disease progression, liver ca development, organoids.)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Lazaridis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States